CLINICAL TRIAL: NCT00802685
Title: Timing of PDA Closure and Respiratory Outcome in Premature Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of availability of IV ibuprofen as of 8/10 due to a manufacturer's recall
Sponsor: University of Miami (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Ilene R.S. Sosenko, M.D., Professor of Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070871
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2013-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent ductus arteriosus; Respiratory outcome
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early ibuprofen (Experimental): Drug: Early ibuprofen
  IBUPROFEN DOSING SCHEDULE: At the diagnosis of PDA, infants randomized to "early treatment" will receive blinded ibuprofen initial dose 10 mg/kg, then two doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Initial therapy will be blinded. This group will then be eligible to receive unblinded, open label ibuprofen for a hemodynamically significant PDA include: SIGNS OF PDA + Presence of significant pulmonary hemorrhage ALONE OR SIGNS OF PDA +: Pulmonary edema, plus a large heart on CXR + one of the following: Hypotension, Respiratory failure (not due to something other than PDA) defined as at least two of the following respirator settings: Need for supplemental O2 > 50%; need IMV >40; need for PIP > 20; or need for HFOV.
  Interventions: Drug: Early ibuprofen
- Late Ibuprofen expectant group (placebo) (Other): Late ibuprofen expectant group (placebo): Ibuprofen schedule: At PDA diagnosis, infants randomized to "late expectant group" will receive blinded placebo. If hemo-dynamically significant PDA develops, infants now receive open label ibuprofen, initial dose of 10 mg/kg, then 2 doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Signs of a hemodynamically significant PDA: Signs of PDA + pulmonary hemorrhage alone or Signs of PDA + Pulmonary edema, plus a large heart on CXR + one of the following: Hypotension, Respiratory failure (due to PDA) defined as at least two of the following respirator settings: Need for supplemental O2 > 50%; need IMV >40; need for PIP > 20; or need for HFOV. Infants who had received placebo will ibuprofen for the first time (thus, "late" ibuprofen or expectant).
  Interventions: Other: Late ibuprofen expectant group (placebo)

INTERVENTIONS:
Drug: Early ibuprofen — IBUPROFEN SCHEDULE: initial dose 10 mg/kg, then 2 doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Initial therapy is blinded. At PDA diagnosis, infants randomized to "early treatment" receive blinded ibuprofen. Infants randomized to "late treatment" receive blinded placebo. Hemodynamically significant PDA criteria: SIGNS OF PDA + pulmonary hemorrhage OR SIGNS OF PDA +: Pulmonary edema, plus a large heart on CXR + one of the following: Hypotension, Respiratory failure (due to PDA) defined as at least two of the following: Need for supplemental O2 > 50%; need IMV >40; need for PIP > 20; or need for HFOV. Once hemodynamically significant PDA criteria met, if echo is positive, infants from both groups can receive open label ibuprofen.
  Arms: early ibuprofen
Other: Late ibuprofen expectant group (placebo) — Drug: Late ibuprofen expectant group (placebo): DOSING SCHEDULE: At PDA diagnosis infants randomized to "late ibuprofen expectant group" will receive blinded placebo. If hemodynamically significant PDA develops, infants now receive open label ibuprofen at an initial dose of 10 mg/kg, then two doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Signs of a hemodynamically significant PDA include: SIGNS OF PDA + pulmonary hemorrhage ALONE OR SIGNS OF PDA +: Pulmonary edema, plus a large heart on CXR + one of the following: Hypotension, Respiratory failure (due PDA) defined as at least 2 of the following settings: Need for supplemental O2 > 50%; need IMV >40; need for PIP > 20; or need for HFOV.
  Arms: Late Ibuprofen expectant group (placebo)

SUMMARY:
The investigators propose the present study with the following aims:

* to determine whether early patent ductus arteriosus (PDA) treatment with ibuprofen treatment at the onset of clinical symptoms is superior to late ibuprofen treatment only when symptoms of a hemodynamically significant PDA are present in the evolution of bronchopulmonary dysplasia (BPD) defined as duration of supplemental oxygen exposure during the first 28 days
* to determine whether early PDA treatment with ibuprofen will be superior to late treatment with ibuprofen in efficacy of PDA closure, need for rescue therapy, need for PDA ligation and incidence of major complications of prematurity.

Hypothesis: Early pharmacologic closure of PDA with ibuprofen will improve respiratory course and reduce BPD as reflected by a reduction in duration of supplemental oxygen during the first 28 days of age vs. late pharmacologic treatment with ibuprofen.

Outcome variables: The primary outcome of this study is the number of days spent on supplemental oxygen by each infant during the first 28 days.

Other outcomes to be determined between groups include:

* Mortality
* Other respiratory variables: total days on supplemental oxygen, days on mechanical ventilation, oxygen dependence at 36 weeks post menstrual age, age at final extubation.
* Other respiratory complications: pneumothorax, pulmonary interstitial emphysema, need for high frequency ventilation, pulmonary hypertension
* Efficacy of PDA closure: number of courses of medication required, need for ligation
* Other neonatal complications: intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), retinopathy of prematurity (ROP), necrotizing enterocolitis (NEC), intestinal perforation, sepsis, renal dysfunction (oliguria, elevated creatinine)
* Time to achieving full enteral feedings, time to regain birth weight, weight at discharge.
* Length of hospital stay

DETAILED DESCRIPTION:
Study terminated when intravenous (IV) ibuprofen withdrawn for both clinical and research use.

ELIGIBILITY:
Inclusion Criteria:

* Inborn patients at JHS hospitals (admitted to the NICU at JMH within the first 72 hrs of age
* BW 500-1250 grams
* 23-32 wks gestational age
* > 1d but < 14d of age.

Exclusion Criteria:

* Major congenital malformations
* Proven sepsis (positive blood culture)
* Contraindications to the use of Ibuprofen or Indomethacin
* Terminal condition, not expected to survive beyond 48 h
* Infants born excessively SGA(3 S.D. below the mean for GA)
* Infants with initial PDA presentation that is hemodynamically significant

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilene RS Sosenko, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital/Holtz Children's Center, Miami, Florida, United States

REFERENCES:
- [Derived] Sosenko IR, Fajardo MF, Claure N, Bancalari E. Timing of patent ductus arteriosus treatment and respiratory outcome in premature infants: a double-blind randomized controlled trial. J Pediatr. 2012 Jun;160(6):929-35.e1. doi: 10.1016/j.jpeds.2011.12.031. Epub 2012 Jan 28. PMID 22284563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initiated on 01/02/08; the final patient was recruited on 7/26/10. Patients were enrolled at Jackson Memorial Hospital. Study was terminated early due to lack of availability of IV ibuprofen due to manufacturer's recall.
Pre-assignment Details: 179 subjects had consents obtained. Of these, 6 consents were withdrawn and 68 enrolled subjects were not randomized because they met exclusion criterion before randomization: hemodynamically significant PDA (n=10), absence of PDA (n=55) and other reasons (n=3).
  Therefore 105 enrolled subjects were randomized into 1 of 2 treatment arms.
Groups:
- Early Ibuprofen: Drug: Early ibuprofen IBUPROFEN DOSING SCHEDULE: At the diagnosis of PDA, infants randomized to "early treatment" will receive blinded ibuprofen initial dose 10 mg/kg, then two doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Initial therapy will be blinded. This group will then be eligible to receive unblended, open label ibuprofen for a hemodynamically significant PDA include: SIGNS OF PDA + Presence of significant pulmonary hemorrhage ALONE OR SIGNS OF PDA +: Pulmonary edema, plus a large heart on CXR + one of the following: Hypotension, Respiratory failure (not due to something other than PDA) defined as at least two of the following respirator settings: Need for supplemental O2 > 50%; need IMV >40; need for PIP > 20; or need for HFOV.
  Early ibuprofen : IBUPROFEN DOSING SCHEDULE: initial dose 10 mg/kg, then two doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Initial therapy will be blinded. At the diagnosis of PDA, infants randomized to "early treatment" w
- Late Ibuprofen Expectant Group: Drug: Late ibuprofen expectant group
  IBUPROFEN DOSING SCHEDULE: At the diagnosis of PDA, infants randomized to "late ibuprofen expectant group" will receive blinded placebo. If criteria of a hemodynamically significant PDA develop, infants from this group can now receive open label ibuprofen at an initial dose of 10 mg/kg, then two doses 5 mg/kg each, after 24 and 48 h, slow IV infusion. Signs of a hemodynamically significant PDA include: SIGNS OF PDA + Presence of significant pulmonary hemorrhage ALONE OR SIGNS OF PDA +: Pulmonary edema, plus a large heart on CXR + one of the following: Hypotension, Respiratory failure (not due to something other than PDA) defined as at least two of the following respirator settings: Need for supplemental O2 > 50%; need IMV >40; need for PIP > 20; or need for HFOV. Infants who had received placebo will be have ibuprofen for the first time (thus, "late" ibuprofen or expectant).
  Late ibuprofen expectant group : Other: Late Ibuprofen expectant
Period: Overall Study
Arm/Group | Early Ibuprofen | Late Ibuprofen Expectant Group
Started | 54 | 51
Completed | 54 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Ibuprofen | Late Ibuprofen Expectant Group | Total
Number analyzed (Participants) | 54 | 51 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 51 | 105
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 50
  Male | 25 | 30 | 55
Region of Enrollment [Number; unit: participants]
  United States | 54 | 51 | 105

OUTCOME MEASURES:

1. Primary Outcome: Days Spent on Supplemental Oxygen During the First 28 Days.
Time Frame: 28 days of life
Population: The number of participants for analysis was determined from all subjects who completed the study intervention at 28 days of age and had complete data on the primary endpoint of oxygen days during the first 28 days. Analysis was done on intention to treat basis.
Measure: Median (Full Range); unit: days
Arm/Group | Early Ibuprofen | Late Ibuprofen Expectant Group
Number analyzed (Participants) | 54 | 51
days | 21 [7 to 27] | 19 [5 to 26]
Statistical Analysis 1: Comparison: Early Ibuprofen vs Late Ibuprofen Expectant Group; Null hypothesis: Oxygen duration (days) during the first 28 days will be equal between treatment arms; Test type: Superiority or Other; p = 0.858, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4, 95% CI 2-sided [4 to 36], Standard Deviation 8

2. Secondary Outcome: Number of Participants on Oxygen at 36 Weeks Postmenstrual Age
Time Frame: at 36 weeks postmenstrual age
Measure: Number; unit: participants
Arm/Group | Early Ibuprofen | Late Ibuprofen Expectant Group
Number analyzed (Participants) | 54 | 51
participants | 17 [15 to 20] | 16 [15 to 20]
Statistical Analysis 1: Comparison: Early Ibuprofen vs Late Ibuprofen Expectant Group; null hypothesis: The proportion of subjects on O2 at 36 wk PMA will be equal between treatment arms; Test type: Superiority or Other; p = 0.8, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.953, 95% CI 2-sided [0.393 to 2.309]

ADVERSE EVENTS:
Arm/Group | Early Ibuprofen | Late Ibuprofen Expectant Group
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 0/54 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes